CLINICAL TRIAL: NCT02497352
Title: Effects of Flaxseed Supplementation in Metabolic Syndrome
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Principal Investigator, Dr Azita Hekmatdoost, Principal Investigator, National Nutrition and Food Technology Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 765
Record Dates: First submitted 2015-07-10; First posted 2015-07-14 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2014-12

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Linseed Oil

ARMS (2):
- Flaxseed (Experimental): 30 g milled brown flaxseed + lifestyle modification
  Interventions: Dietary Supplement: flaxseed; Behavioral: lifestyle modification
- control (Active Comparator): lifestyle modification including dietary and physical activity recommendation
  Interventions: Behavioral: lifestyle modification

INTERVENTIONS:
Dietary Supplement: flaxseed
  Arms: Flaxseed
Behavioral: lifestyle modification

SUMMARY:
To evaluate the effects of flaxseed supplementation on fasting blood sugar, lipid profile and anthropocentric measurements in subjects with metabolic syndrome, in a randomized, open-labeled, controlled pilot study, 44 subjects with metabolic syndrome will be received 30g/d flaxseed with lifestyle modification or lifestyle modification alone for 12 weeks. Both groups will be advised to follow an energy balanced diet and physical activity recommendations. Parameters related to metabolic syndrome will be measured at the baseline and at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* having three of the following five features: Increased waist circumference (≥102 cm in men and ≥88 cm in women), elevated TG (≥150 mg/dl), reduced HDL-C (≤40 mg/dl in men and ≤50 mg/dl in women), elevated blood pressure (≥130/85 mm Hg or on treatment for hypertension) and elevated glucose (≥100 mg/dl), according to the National Cholesterol Education Program Adult Treatment Panel III report

Exclusion Criteria:

* history of allergy or high consumption of nuts, flaxseed, or sesame seeds
* clinically diagnosed renal, liver, heart, pituitary, thyroid, or psychiatric disorders impairing the patient's ability to provide written informed consent
* history of cardiovascular diseases, cancers, alimentary tract disorders affecting absorption
* pregnancy, lactation, and lack of effective birth control in women of child-bearing potential

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-02; Primary Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Insulin resistance index (HOMA-IR) | 12 weeks
  The homeostatic model assessment (HOMA)